CLINICAL TRIAL: NCT03448094
Title: The Acute and Chronic Effects of Resveratrol Supplementation on Cognitive Function, Gastrointestinal Microbiota and Cerebral Blood Flow: a Double-blind, Placebo-controlled, Parallel-groups Study in Healthy, Overweight Humans.
Brief Title: The Effects of Resveratrol Supplementation on Cognition, Cerebral Blood Flow, Microbiota and Systemic Inflammation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Evolva SA (Industry)
Responsible Party: Principal Investigator, EllenSmith, PhD Researcher, Northumbria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 52P6
Record Dates: First submitted 2018-02-07; First posted 2018-02-27 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Cognitive Function and Mood; Cerebral Blood Flow; Systemic Inflammation; Gut Microbiota; Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Resveratrol

STUDY DESIGN:
Intervention Model Description: Participants will recieve either Resveratrol or Placebo for a period of 3 months.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resveratrol (Experimental): 500mg of Veri-te Resveratrol (consumed as two 250mg tablets, at two timepoints each day).
  Interventions: Dietary Supplement: Resveratrol
- Placebo (Placebo Comparator): Matched placebo capsules (1 capsule consumed at two timepoints each day).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Resveratrol — Participants will consume one of the treatment types daily for a period of three months.
  Other Names: Veri-teTM Resveratrol
  Arms: Resveratrol
Dietary Supplement: Placebo — Participants will consume one of the treatment types daily for a period of three months.
  Arms: Placebo

SUMMARY:
Previous research shows that a diet high in fat has harmful effects on gut health. This increases the chance of developing obesity-related diseases (such as type 2 diabetes) and disrupts cognition and mood.

Research has suggested that gut health can be improved by taking certain supplements, including resveratrol (a polyphenol found primarily in red grape skins). Resveratrol has also been shown to improve brain blood flow and possibly brain function - however, there is limited research studying this.

This study will investigate the effects of 12 weeks daily consumption of resveratrol on cognitive function, cerebral blood flow, gut microbiota and systemic inflammation in overweight and obese healthy adults.

DETAILED DESCRIPTION:
Each participant will be required to attend the laboratory on four occasions. The first of these will be an initial screening/training visit, this will take place in the afternoon and last 3 hours in total. During the initial visit participants will be asked to provide written informed consent. They will provide lifestyle and demographic data and screened regards to physical health (height, weight, blood pressure, waist to hip ratio). They will then be trained on the computerised cognitive and mood tasks. At the end of the appointment they will be provided with a food diary and a stool sample collection kit.

Study days 1 and 2 (12 weeks apart) :

Participants will arrive at the laboratory at 8.00am having fasted from 8pm the previous evening, avoided caffeinated products for 18 hours, alcohol and over the counter medication for 24 hours and oral antihistamines for 48 hours prior to the session commencing. They will also bring with them their completed food diary and stool sample.

Participants will provide a blood sample and then will be given a standardised breakfast of x2 slices of white toast with butter and a decaf tea or coffee. They will also provide a urine sample. Participants will then complete a computerised cognitive assessment (~1 hour in length), followed by measurements of blood pressure and heart rate. Participants in the sub-sample who will also provide brain (cerebral) blood flow data, will then have the quantitative near-infrared spectroscopy (qNIRS) headband fitted across the forehead and a 5 minute baseline measure will be recorded.

Following this the participants will consume their treatment for the day, followed by a short break and then will complete the second cognitive assessment. The qNIRS participants will again provide brain blood flow data and following that will be provided with a standardised lunch (cheese sandwich, ready salted crisps and a custard pot). Participants will complete their final cognitive assessment and will then provide a second blood sample.

At the end of the first study day participants will be provided with their treatment and treatment diary, they will be instructed to take one tablet twice a day (with breakfast and dinner). Both study days will be identical and will take place 84 days (+/- 5 days) apart.

Participants are also required to attend a short treatment exchange visit during Week 6 (5 minutes).

ELIGIBILITY:
Inclusion Criteria:

* Interested in taking part in the study
* Healthy
* Aged 35-60 years (inclusive)
* Have a BMI of between 25-39.9
* Willing to consume your normal diet during the 12 week supplementation period

Exclusion Criteria:

You should not take part if you:

* Are aged under 35 or over 60
* Have a Body Mass Index (BMI) lower than 25 or higher than 39.9.
* Have taken antibiotics (including pre- and pro-biotic supplements/drinks) during the previous 8 weeks
* Have irregular bowel movements (less than 1 per day)
* Have any pre-existing medical conditions/illness with some exceptions - please check with the researcher
* Have type 1 or type 2 diabetes
* Are currently taking prescription medications with some exceptions- please check with the researcher
* Have a visual impairment that cannot be corrected by glasses or contact lenses, including colour blindness.
* English is not your first language or your English proficiency is not equivalent to the International English language test system (IELTS) band 6 or above
* Have any learning difficulties or dyslexia
* Currently suffer from frequent migraines that require medication (>1 per month)
* Have any food allergies, intolerances or sensitivities
* Have high blood pressure (systolic over 159 mm Hg or diastolic over 99 mm Hg)
* Smoke
* Have a history of alcohol or drug abuse
* Are pregnant, seeking to become pregnant or lactating
* Are unable to complete all of the study assessments
* Are currently participating in any other clinical or nutritional intervention study, or have done within the past 4 weeks
* Have any health condition that would prevent fulfilment of the study requirements
* Have habitually used supplements within the last month (defined as more than 3 consecutive days or 4 days in total)
* Have an excessive caffeine intake (>500mg per day) - equivalent to 5/6 cups of coffee/8 cups of tea per day or equivalent from other sources
* Consume more than 5 portions of fruit or vegetables per day
* Any sleep disturbances or take sleep aid medication
* Have any known active infections
* You have or may think you are at risk of having syphilis, hepatitis, the Human T - lymphotropic virus or the Human Immunodeficiency Virus?
* You have ever had breast cancer and/or a mastectomy
* You have haemophilia or any similar clotting disorder
* Do not have a bank account (required for payment)

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2019-07-13 (Actual); Study Completion 2019-07-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline cognitive (memory) performance at 45 minutes, 240 minutes and 12 weeks post dose | 45 minutes, 240 minutes, 12 weeks
  Memory performance will be assessed using a computerised cognitive battery (administered using COMPASS cognitive assessment program). Memory will be assessed using 3 global measures (Working memory, speed of memory and episodic memory). The global measures are created by taking data from several tasks targeting that cognitive domain. Working memory: a combined accuracy score (% correct) from the tasks: numeric working memory (NWM), serial 3's subtractions (SS3), serial 7's subtractions (SS7) and rapid visual information processing (RVIP). Speed of memory: a combined speed score (msecs) from tasks NWM, delayed name to face recall, delayed picture recognition and delayed word recognition. Episodic memory: a combined accuracy score (% correct) from tasks immediate word recall, delayed word recall, delayed name to face recall, delayed picture recognition, delayed word recognition.
Change from baseline cognitive (Attention) performance at 45 minutes, 240 minutes and 12 weeks post dose | 45 minutes, 240 minutes, 12 weeks
  Attention performance will be assessed using a computerised cognitive battery (administered using COMPASS cognitive assessment program). Attention will be assessed using 2 global measures (Accuracy of Attention and Speed of Attention). Accuracy of Attention: accuracy score (% correct) from choice reaction time task. Speed of attention: speed score (msecs) taken from choice reaction time task.
Gut microbiota | 12 weeks
  Changes in gut microbiota communities, quantified using 16S ribosomal ribonucleic acid (rRNA) gene community analysis.
Change from baseline systemic inflammatory cytokines | 5 hours, 12 weeks
  Inflammatory cytokines (including C-reactive protein and Interleukin-6) will be measured in plasma using ELISA analysis, in association with other endpoints including resveratrol metabolites.
Change from baseline urinary and plasma metabolome | 12 weeks
  Changes in plasma and urinary metabolome will be profiled using a Thermo Q-Exactive liquid chromatography/mass spectrometry spectrometer and data analysed using Progenesis QI.
Change from baseline total haemoglobin cerebral blood flow (CBF) measurement | 115-190 minutes, 12 weeks
  CBF of the frontal cortex measured using quantitative near infrared spectroscopy (q-NIRS).
Change from baseline deoxygenated haemoglobin CBF measurement | 115-190 minutes, 12 weeks
  CBF of the frontal cortex measured using qNIRS.
Change from baseline oxygen saturation CBF measurement | 115-190 minutes, 12 weeks
  CBF of the frontal cortex measured using qNIRS.

SECONDARY OUTCOMES:
Change from baseline Blood Pressure | 45 minutes, 240 minutes, 12 weeks
  Systolic and diastolic blood pressure will be taken after each cognitive assessment (measured in mm Hg).
Change from baseline Heart Rate | 45 minutes, 240 minutes, 12 weeks
  Heart rate will be measured after each cognitive assessment (measured in BPM).
Change from baseline subjective mood score | 240 minutes, 12 weeks
  Subjective mood scores will be measured using the Profile of Mood scale. The questionnaire includes 65 items and participants rate their mood on a scale of 0-4 (not at all - extremely). These scores are collapsed into 6 mood outcomes (Tension, depression, anger, vigour, fatigue and confusion) and a total mood disturbance score.
Weight change and BMI | 12 weeks
  Change in weight and BMI between visits

CONTACTS AND LOCATIONS:
Overall Officials: Emma Wightman, Dr, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No